CLINICAL TRIAL: NCT02650713
Title: An Open-Label, Multicenter, Dose Escalation and Expansion Phase Ib Study to Evaluate the Safety, Pharmacokinetics, and Therapeutic Activity of RO6958688 in Combination With Atezolizumab in Patients With Locally Advanced and/or Metastatic CEA-Positive Solid Tumors
Brief Title: A Study of the Safety, Pharmacokinetics, and Therapeutic Activity of RO6958688 in Combination With Atezolizumab in Participants With Locally Advanced and/or Metastatic Carcinoembryonic Antigen (CEA)-Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WP29945; RG7802 (Other: Roche); 2015-003771-30 (EudraCT Number)
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose-Escalation (Part IA): RO6958688 + Atezolizumab (Experimental): Participants will receive RO6958688 weekly (QW) at escalating doses starting at 5 mg, in combination with a fixed dose (1200 mg) of atezolizumab every 3 weeks (Q3W). RO6958688 dosage will not exceed the MTD if defined in the BP29541 study.
  Interventions: Drug: Atezolizumab; Drug: RO6958688
- Dose/Schedule Finding (Part IB): RO6958688 + Atezolizumab (Experimental): Part IB will explore different RO6958688 administration schedules in combination with atezolizumab, consisting of:
  Cohort A: will compare the QW vs Q3W dosing schedules at a flat dose of RO6958688.
  Step Up dosing schedules: RO6958688 dose will start at 40 mg and increase with each administration up to the MTD or 1200 mg, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: RO6958688

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose of 1200 milligrams (mg) by intravenous (IV) infusion.
  Other Names: Tecentriq
Drug: RO6958688 — RO6958688 is administered by IV infusion
  In Part IA: RO6958688 is administered weekly (QW) on days 1,8 and 15 of each 21-day cycle.
  In Part 1b: RO6958688 is administered weekly (QW) or every 3 weeks (Q3W). Cohort A: RO6958688 starting dose will be 100 mg either QW or Q3W.
  Step Up dose cohorts: RO6958688 starting dose will be 40mg and increase with each administration up to the MTD or 1200 mg whichever is lower.

SUMMARY:
This is an open-label, multicenter, dose-escalation and expansion Phase Ib clinical study of RO6958688 in combination with atezolizumab. Part I of the study is subdivided into parts IA and IB. Part IA is dose escalation with a starting dose of 5 mg of RO6958688 given QW (once a week) and a fixed, flat dose of 1200 mg given Q3W (every 3 weeks) of atezolizumab, to evaluate the safety and determine the MTD of RO6958688 in combination with atezolizumab. Part IB is a dose/schedule finding part that will explore different administration schedules of RO6958688 in combination with atezolizumab (1200 mg Q3W) to establish the appropriate dose/schedule of RO6958688 in combination with atezolizumab.

ELIGIBILITY:
Inclusion Criteria

* Confirmed locally advanced and/or metastatic solid tumor, with at least one tumor lesion of accessible non-critical location to biopsy, in participants who have progressed on a standard therapy, are intolerant to standard therapy, and/or are non-amenable to standard therapy
* Radiologically measurable and clinically evaluable disease (as per RECIST v1.1)
* Life expectancy (in the opinion of the investigator) of at least 12 weeks and lactate dehydrogenase (LDH) levels </= 2.5 ULN (upper limit of normal)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade </= 1 or returned to baseline except alopecia (any grade) and Grade 2 peripheral neuropathy
* Adequate hematological, liver, and renal function
* Negative serum pregnancy test within 7 days prior to study treatment in premenopausal women and women </= 2 years after start of menopause (menopause is defined as amenorrhea for more than 2 years)
* Participants must agree to remain abstinent or be willing to use effective methods of contraception as defined in the protocol
* Participants with non-colorectal cancer should have confirmed CEA expression in tumor tissue. For colorectal cancer (CRC), the CEA assessment should be performed but the result is not required for participant selection

Exclusion Criteria

* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 2 weeks prior to enrollment
* Leptomeningeal disease
* Participants with paraspinal, paratracheal, and mediastinal pathological lesions larger than 2 cm unless they are previously irradiated
* Malignancies within 5 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome
* Significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results
* Uncontrolled hypertension, unstable angina, congestive heart failure (CHF), serious cardiac arrhythmia requiring treatment history of myocardial infarction within 6 months of enrollment
* Administration of a live, attenuated vaccine within 28 days before Cycle 1 Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Human Inmmunodeficiency Virus (HIV), active Hepatitis B or Hepatitis C (HCV)
* Severe infections within 28 days prior to Cycle 1 Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia or active tuberculosis
* Received oral or intravenous (IV) antibiotics within 14 days prior to Day 1
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Major surgery or significant traumatic injury less than 28 days prior to Cycle 1 Day 1 (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Known history of autoimmune disease as defined in the protocol
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis (including drug induced) on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Participants with bilateral lung lesions and dyspnea and/or oxygen saturation level (SaO2) less than 92% (at rest, room air and exertion) or participants with lobectomy or pneumonectomy with lung metastases in the remaining lung and either dyspnea or SaO2 less than 92% (at rest, room air and exertion) at baseline
* Pregnant or breast-feeding
* Known hypersensitivity to any of the components of RO6958688 and atezolizumab; hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Investigational therapy (defined as treatment for which there is no regulatory authority approved indication) or last dose of prior immunotherapies within 28 days prior to Cycle 1 Day 1. Participants previously treated with anti-programmed death-ligand 1 (PD-L1), or anti-PD-1 are excluded
* Last dose of any approved anti-cancer therapy within 28 days prior to the first RO6958688 infusion
* Prior systemic corticosteroids greater than 10mg prednisone (or equivalent) within 14 days of Cycle 1 Day 1. Inhaled and/or topical steroids are permitted
* Expected need for regular immunosuppressive therapy
* Radiotherapy within the last 28 days before Cycle 1 Day 1 with the exception of limited-field palliative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Baseline up to 60 months
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Day 1 up to Day 21
Maximum-Tolerated Dose (MTD) of RO6958688 | Part IA: Day 1 up to Day 21; Part IB Step-up Cohorts: Day 1 up to Day 7 after each dose escalation
Recommended Phase II Dose (RP2D) of RO6958688 | Day 1 up to 60 months

SECONDARY OUTCOMES:
Pharmacokinetic (PK): Area Under the Concentration-Time Curve (AUC) of RO6958688 | Baseline up to 60 months
PK: Volume of Distribution at Steady State (Vss) of RO6958688 | Baseline up to 60 months
PK: Maximum Serum Concentration (Cmax) of RO6958688 | Baseline up to 60 months
PK: Clearance (CL) of RO6958688 | Baseline up to 60 months
PK: AUC of Atezolizumab | Baseline up to 60 months
PK: Vss of Atezolizumab | Baseline up to 60 months
PK: Cmax of Atezolizumab | Baseline up to 60 months
PK: CL of Atezolizumab | Baseline up to 60 months
Pharmacodynamics: Immune Cell Numbers as Assessed using Flow Cytometry | Pre-infusion (1 hour before infusion start) on Day 1 of Cycles 1, 2, 3, 6; Cycle 1 Days 2 and 8 (cycle length=21 days)
Percentage of Participants with Objective Response (Partial Response [PR] or Complete Response [CR] as Assessed Using Response Evaluation Criteria in Solid Tumors [RECIST]) | Baseline up to 60 months
  Assessed at screening and after the start of treatment every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or treatment discontinuation.
Percentage of Participants with Disease Control (PR, CR, or Stable Disease [SD]) as Assessed Using RECIST | Baseline up to 60 months
  Assessed at screening and after the start of treatment every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or treatment discontinuation.
Percentage of Participants with Stable Disease (SD) as Assessed Using RECIST | Baseline up to 60 months
  Assessed at screening and after the start of treatment every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or treatment discontinuation.
Duration of Response (DOR) as Assessed Using RECIST | From initial objective response (PR or CR to the first disease progression or death from any cause (up to 60 months)
  Assessed at screening and after the start of treatment every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or treatment discontinuation.
Progression-Free Survival (PFS) according to RECIST V1.1 | From first study treatment to the first occurrence of objective disease progression or death from any cause (up to 60 months)
  Assessed at screening and after the start of treatment every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or treatment discontinuation.
Overall Survival (OS) | From first study treatment to death from any cause (up to 60 months)
  Assessed at screening and after the start of treatment every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or treatment discontinuation.
Best Overall Response (BOR) | Baseline up to 60 months
  Assessed at screening and after the start of treatment every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- United States (11):
  - UCLA Cancer Center, Santa Monica, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - University Of Colorado, Aurora, Colorado
  - Smilow Cancer Hospital at Yale- New Haven Oncology Investigational Drug Pharmacy, New Haven, Connecticut
  - Dana Farber Can Ins, Boston, Massachusetts
  - Columbia Univ Med Ctr, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Cancer Center, Germantown, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- France (2):
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - IRCCS IST. Tumori Fondaz. Pascale; S.C. Oncologia Medica,Melanoma,Immunoterapia E Terapie Innovative, Napoli, Campania
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
- Antoni Van Leeuwenhoek Ziekenhuis; Gastro-Enterologie, Amsterdam, Netherlands
- Spain (6):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid

REFERENCES:
- [Derived] Martinez-Sabadell A, Morancho B, Rius Ruiz I, Roman Alonso M, Ovejero Romero P, Escorihuela M, Chicote I, Palmer HG, Nonell L, Alemany-Chavarria M, Klein C, Bacac M, Arribas J, Arenas EJ. The target antigen determines the mechanism of acquired resistance to T cell-based therapies. Cell Rep. 2022 Oct 18;41(3):111430. doi: 10.1016/j.celrep.2022.111430. PMID 36261015